CLINICAL TRIAL: NCT05032196
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled, Phase 1b/2a Study of WVE-003 Administered Intrathecally in Patients With Huntington's Disease (SELECT-HD)
Brief Title: Study of WVE-003 in Patients With Huntington's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: WVE-003-001
Record Dates: First submitted 2021-08-18; First posted 2021-09-02 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — Sagittal Abdominal Diameter

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- SAD: Pooled Placebo (Placebo Comparator): Placebo
  Interventions: Drug: SAD: Pooled Placebo
- SAD: 30mg WVE-003 (Experimental): Single Ascending Dose - 30mg WVE-003
  Interventions: Drug: SAD: 30mg WVE-003
- SAD: 60mg WVE-003 (Experimental): Single Ascending Dose - 60mg WVE-003
  Interventions: Drug: SAD: 60mg WVE-003
- SAD: 90mg WVE-003 (Experimental): Single Ascending Dose - 90mg WVE-003
  Interventions: Drug: SAD: 90mg WVE-003
- MD: Placebo (Placebo Comparator): Placebo
  Interventions: Drug: MD: Placebo
- MD: 30mg WVE-003 (Experimental): Multiple Dose - 30mg WVE-003
  Interventions: Drug: MD: 30mg WVE-003

INTERVENTIONS:
Drug: SAD: 30mg WVE-003 — Single ascending dose of 30mg WVE-003, an allele-selective stereopure antisense oligonucleotide (ASO)
  Arms: SAD: 30mg WVE-003
Drug: SAD: 60mg WVE-003 — Single ascending dose of 60mg WVE-003, an allele-selective stereopure antisense oligonucleotide (ASO)
  Arms: SAD: 60mg WVE-003
Drug: SAD: 90mg WVE-003 — Single ascending dose of 90mg WVE-003, an allele-selective stereopure antisense oligonucleotide (ASO)
  Arms: SAD: 90mg WVE-003
Drug: SAD: Pooled Placebo — Single dose of placebo
  Arms: SAD: Pooled Placebo
Drug: MD: 30mg WVE-003 — Three doses of 30mg WVE-003 Q8WK an allele-selective stereopure, antisense oligonucleotide (ASO)
  Arms: MD: 30mg WVE-003
Drug: MD: Placebo — Three doses of placebo Q8WK
  Arms: MD: Placebo

SUMMARY:
This is a Phase 1b/2a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of WVE-003 in adult patients with early-manifest HD who carry the targeted single nucleotide polymorphism (SNP) - SNP3.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of the A variant of SNP3 on the same allele as the pathogenic CAG triplet expansion
2. Ambulatory, male or female patients aged ≥25 to ≤60 years
3. Clinical diagnostic motor features of HD, defined as Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Score = 4
4. UHDRS Total Functional Capacity Scores ≥9 and ≤13

Exclusion Criteria:

1. Malignancy or received treatment for malignancy, other than treated basal cell or squamous cell carcinoma of the skin, within the previous 5 years
2. Received any other study drug, including an investigational oligonucleotide, within the past 1 year or 5 half-lives of the drug, whichever is longer, with the exception of the following:

   a. Received WVE-120101 or WVE-120102 within the last 3 months
3. Implantable CNS device that may interfere with ability to administer study drug via lumbar puncture or undergo MRI scan
4. Inability to undergo brain MRI (with or without sedation)
5. Bone, spine, bleeding, or other disorder that exposes the patient to risk of injury or unsuccessful lumbar puncture
6. Previously received tominersen

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Wave Life Sciences
Locations (23):
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Monash Health, Clayton, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre Hospitalier de l-Universite de Montreal, Montreal, Quebec
- Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Hopital Henri Mondor - Hospital, Créteil
  - Institut du Cerveau et de la Moelle Epiniere, Paris
- Germany (3):
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - George-Huntington-Institut GmbH, Münster
  - kbo-Isar-Amper-Klinikum Taufkirchen (Vils), Taufkirchen
- Centro Ricerche Cliniche Di Verona, Verona, Italy
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
- Poland (2):
  - Szpital Sw. Wojciecha, Gdansk
  - Instytut Psychiatrii I Neurologii, Warsaw
- Spain (2):
  - Hospital de la Sanata Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
- United Kingdom (4):
  - Royal Devon and Exeter Hospital NHS Trust, Exeter, Devon
  - Royal Hospital for Children, Pharmacy Aseptic Unit, Glasgow, Glasgow City
  - Cardiff University, Schools of Medicine and Biosciences, Cardiff, Wales
  - Royal Liverpool University Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iwamoto N, Liu Y, Frank-Kamenetsky M, Maguire A, Tseng WC, Taborn K, Kothari N, Akhtar A, Bowman K, Shelke JD, Lamattina A, Hu XS, Jang HG, Kandasamy P, Liu F, Longo K, Looby R, Meena, Metterville J, Pan Q, Purcell-Estabrook E, Shimizu M, Prakasha PS, Standley S, Upadhyay H, Yang H, Yin Y, Zhao A, Francis C, Byrne M, Dale E, Verdine GL, Vargeese C. Preclinical evaluation of stereopure antisense oligonucleotides for allele-selective lowering of mutant HTT. Mol Ther Nucleic Acids. 2024 Jun 11;35(3):102246. doi: 10.1016/j.omtn.2024.102246. eCollection 2024 Sep 10. PMID 39027419
- [Derived] Estevez-Fraga C, Tabrizi SJ, Wild EJ. Huntington's Disease Clinical Trials Corner: November 2022. J Huntingtons Dis. 2022;11(4):351-367. doi: 10.3233/JHD-229006. PMID 36463457

RESULTS

PARTICIPANT FLOW:
Groups:
- SAD: Pooled Placebo: SAD: Single dose of placebo.
- SAD: 30mg WVE-003*: SAD: Single ascending dose of 30mg WVE-003. *
- SAD: 60mg WVE-003*: SAD: Single ascending dose of 60mg WVE-003. *
- SAD: 90mg WVE-003: SAD: Single ascending dose of 90mg WVE-003.
- MD: Placebo: MD: 3 doses of placebo Q8W. 7 Pts from Period 1 rolled over into Period 2.
- MD: 30mg WVE-003: MD: 3 doses of 30mg WVE-003 Q8W. 16 Pts rolled over from Period 1 into Period 2.
Period: Period 1 (Single Ascending Dose)
Arm/Group | SAD: Pooled Placebo | SAD: 30mg WVE-003* | SAD: 60mg WVE-003* | SAD: 90mg WVE-003 | MD: Placebo | MD: 30mg WVE-003
Started | 16 | 12 | 11 | 8 | 0 | 0
Completed (1 Pt was randomized to WVE-003 60mg SAD group but received 30mg instead. This Pt is counted in the 30mg arm, but appears in the 60mg arm in the study flow diagram.) | 16 | 11 | 11 | 7 | 0 | 0
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 2 (Multidose)
Arm/Group | SAD: Pooled Placebo | SAD: 30mg WVE-003* | SAD: 60mg WVE-003* | SAD: 90mg WVE-003 | MD: Placebo | MD: 30mg WVE-003
Started | 0 | 0 | 0 | 0 | 7 | 16
Treated | 0 | 0 | 0 | 0 | 7 | 16
Completed | 0 | 0 | 0 | 0 | 6 | 16
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MD: 30mg WVE-003: Multiple Dose - 30mg WVE-003
  MD: 30mg WVE-003: Three doses of 30mg WVE-003 Q8WK an allele-selective stereopure antisense oligonucleotide (ASO
- Total: Total of all reporting groups
Arm/Group | SAD: Pooled Placebo | SAD: 30mg WVE-003 | SAD: 60mg WVE-003 | SAD: 90mg WVE-003 | MD: Placebo | MD: 30mg WVE-003 | Total
Number analyzed (Participants) | 16 | 13 | 10 | 8 | 7 | 16 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 47 participants were enrolled into Period 1, and of those 23 participants were rolled over into Period 2.
  years
    Period 1: number analyzed (Participants) | 16 | 13 | 10 | 8 | 0 | 0 | 47
    Period 1 | 45.5 (7.4) | 47.8 (9.2) | 43.9 (8.6) | 49.6 (5.3) |  |  | 46.5 (7.9)
    Period 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 16 | 23
    Period 2 |  |  |  |  | 45.6 (8.3) | 47.8 (8.3) | 47.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 47 participants were enrolled into Period 1, and of those 23 participants were rolled over into Period 2.
  Participants
    Period 1: number analyzed (Participants) | 16 | 13 | 10 | 8 | 0 | 0 | 47
    Period 1: Female | 6 | 6 | 3 | 3 |  |  | 18
    Period 1: Male | 10 | 7 | 7 | 5 |  |  | 29
    Period 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 16 | 23
    Period 2: Female |  |  |  |  | 2 | 5 | 7
    Period 2: Male |  |  |  |  | 5 | 11 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 47 participants were enrolled into Period 1, and of those 23 participants were rolled over into Period 2.
  Participants
    Period 1: number analyzed (Participants) | 16 | 13 | 10 | 8 | 0 | 0 | 47
    Period 1: Hispanic or Latino | 1 | 0 | 0 | 0 |  |  | 1
    Period 1: Not Hispanic or Latino | 15 | 13 | 10 | 8 |  |  | 46
    Period 1: Unknown or Not Reported | 0 | 0 | 0 | 0 |  |  | 0
    Period 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 16 | 23
    Period 2: Hispanic or Latino |  |  |  |  | 1 | 0 | 1
    Period 2: Not Hispanic or Latino |  |  |  |  | 6 | 16 | 22
    Period 2: Unknown or Not Reported |  |  |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 47 participants were enrolled into Period 1, and of those 23 participants were rolled over into Period 2.
  Participants
    Period 1: number analyzed (Participants) | 16 | 13 | 10 | 8 | 0 | 0 | 47
    Period 1: American Indian or Alaska Native | 0 | 0 | 0 | 0 |  |  | 0
    Period 1: Asian | 0 | 0 | 0 | 0 |  |  | 0
    Period 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  |  | 0
    Period 1: Black or African American | 0 | 0 | 0 | 0 |  |  | 0
    Period 1: White | 16 | 13 | 10 | 8 |  |  | 47
    Period 1: More than one race | 0 | 0 | 0 | 0 |  |  | 0
    Period 1: Unknown or Not Reported | 0 | 0 | 0 | 0 |  |  | 0
    Period 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 16 | 23
    Period 2: American Indian or Alaska Native |  |  |  |  | 0 | 0 | 0
    Period 2: Asian |  |  |  |  | 0 | 0 | 0
    Period 2: Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 | 0 | 0
    Period 2: Black or African American |  |  |  |  | 7 | 16 | 23
    Period 2: White |  |  |  |  | 0 | 0 | 0
    Period 2: More than one race |  |  |  |  | 0 | 0 | 0
    Period 2: Unknown or Not Reported |  |  |  |  | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety: Proportion of Patients With Treatment Emergent Adverse Events (TEAEs) Related to Study Drug
Description: The primary outcome for this study was safety and is reported as the proportion of patients with TEAEs related to study drug.
Time Frame: Day 1 through Week 24 (single ascending dose Period 1); Day 1 through Week 28 (multi dose Period 2)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD: Pooled Placebo | SAD: 30mg WVE-003 | SAD: 60mg WVE-003 | SAD: 90mg WVE-003 | MD: Placebo | MD: 30mg WVE-003
Number analyzed (Participants) | 16 | 13 | 10 | 8 | 7 | 16
Participants | 2 | 1 | 3 | 3 | 0 | 8

2. Secondary Outcome: Pharmacokinetics of WVE-003 in Plasma
Description: Parameter analyzed: AUC0-6 = area under the concentration-time curve from time 0 to 6 hrs
Time Frame: Day 1 (single ascending dose Period 1); Day 1 and Day 113 (multi dose Period 2)
Population: Please note that the PK analysis only includes participants treated with WVE-003 (all placebo participants have been set as '0').
Measure: Mean (Standard Deviation); unit: AUC 0-6 (hr*ng/mL)
Arm/Group | SAD: 30mg WVE-003 | SAD: 60mg WVE-003 | SAD: 90mg WVE-003 | MD: 30mg WVE-003
Number analyzed (Participants) | 13 | 10 | 8 | 16
AUC 0-6 (hr*ng/mL)
  D1: AUC 0-6 (hr*ng/mL) | 1000 (702) | 2310 (3090) | 3890 (2900) | 822 (409)
  D113: AUC 0-6 (hr*ng/mL): number analyzed (Participants) | 0 | 0 | 0 | 16
  D113: AUC 0-6 (hr*ng/mL) |  |  |  | 698 (432)

3. Secondary Outcome: Pharmacokinetics of WVE-003 in Plasma
Description: Parameter analyzed: Cmax = maximum observed concentration.
Time Frame: Day 1 (single ascending dose Period 1); Day 1 and Day 113 (multi dose Period 2)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Cmax (ng/mL)
Arm/Group | SAD: 30mg WVE-003 | SAD: 60mg WVE-003 | SAD: 90mg WVE-003 | MD: 30mg WVE-003
Number analyzed (Participants) | 13 | 10 | 8 | 16
Cmax (ng/mL)
  D1: Cmax (ng/mL) | 240 (168) | 601 (774) | 1061 (942) | 186 (106)
  D113: Cmax (ng/mL): number analyzed (Participants) | 0 | 0 | 0 | 16
  D113: Cmax (ng/mL) |  |  |  | 157 (97.3)

4. Secondary Outcome: Concentration of WVE-003 in Cerebrospinal Fluid (CSF)
Description: WVE-003 concentration in cerebrospinal fluid (CSF) is reported in ng/mL.
Time Frame: 28 days post-dose during Period 1 (P1:Day29); 28 days post last dose during Period 2 (P2: Day141)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAD: 30mg WVE-003 | SAD: 60mg WVE-003 | SAD: 90mg WVE-003 | MD: 30mg WVE-003
Number analyzed (Participants) | 13 | 10 | 8 | 16
ng/mL | 3.6405 (1.6133) | 5.5346 (2.8402) | 7.0983 (3.1335) | 4.2903 (1.9722)

ADVERSE EVENTS:
Time Frame: Day 1 through Week 24 (single ascending dose Period 1); Day 1 through Week 28 (multi dose Period 2)
Description: This study protocol collected all treatment-emergent adverse events and serious adverse events, whether they were treatment related or not. 5 months after a patient completed their final safety visit, an SAE was reported that sponsor assessed to be not-related to WVE-003.
Groups:
- SAD: 30mg WVE-003: Single Ascending Dose - 30mg WVE-003
  SAD: 30mg WVE-003: Single ascending dose of 30mg WVE-003, a stereopure antisense oligonucleotide (ASO)
- SAD: 60mg WVE-003: Single Ascending Dose - 60mg WVE-003
  SAD: 60mg WVE-003: Single ascending dose of 60mg WVE-003, a stereopure antisense oligonucleotide (ASO)
- SAD: 90mg WVE-003: Single Ascending Dose - 90mg WVE-003
  SAD: 90mg WVE-003: Single ascending dose of 90mg WVE-003, a stereopure antisense oligonucleotide (ASO)
- MD: 30mg WVE-003: Multiple Dose - 30mg WVE-003
  MD: 30mg WVE-003: Three doses of 30mg WVE-003 Q8WK a stereopure antisense oligonucleotide (ASO
Arm/Group | SAD: Pooled Placebo | SAD: 30mg WVE-003 | SAD: 60mg WVE-003 | SAD: 90mg WVE-003 | MD: Placebo | MD: 30mg WVE-003
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13 | 0/10 | 0/8 | 0/7 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/13 | 1/10 | 0/8 | 0/7 | 0/16
Other Adverse Events (participants affected / at risk) | 13/16 | 9/13 | 8/10 | 8/8 | 7/7 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAD: Pooled Placebo (N=16) | SAD: 30mg WVE-003 (N=13) | SAD: 60mg WVE-003 (N=10) | SAD: 90mg WVE-003 (N=8) | MD: Placebo (N=7) | MD: 30mg WVE-003 (N=16)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAD: Pooled Placebo (N=16) | SAD: 30mg WVE-003 (N=13) | SAD: 60mg WVE-003 (N=10) | SAD: 90mg WVE-003 (N=8) | MD: Placebo (N=7) | MD: 30mg WVE-003 (N=16)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 0 | 1 | 1 | 2
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 3 | 2 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 2 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 1 | 0
CSF white blood cell count increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
CSF protein increased (Investigations) | 0 | 2 | 1 | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 1 | 2 | 0
Headache (Nervous system disorders) | 6 | 4 | 2 | 4 | 3 | 4
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleocytosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Intracranial hypotension (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Puncture site pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infected seroma (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
CSF red blood cell count positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Compulsions (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT05032196/Prot_SAP_000.pdf